CLINICAL TRIAL: NCT06403423
Title: Screening for Infra-renal Abdominal Aortic Aneurysms in 65-year-old Men in Inland, Norway
Brief Title: Screening for Aortic Aneurysms in Inland Norway
Acronym: NOR-AORTA
Status: Enrolling by invitation | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Other Study IDs: SI-150503
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Aortic Aneurysm; Erectile Dysfunction; Quality of Life
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with AAA: 65-year old men in Inland, Norway will be invited by mail to a screening. Patients with detected aneurysm will be followed over time with blood samples and questionnaires in addition to ultrasound measurement of the diameter of the infrarenal abdominal aortic aneurysm.
- Control group (no AAA): 65-year old men in Inland, Norway will be invited by mail to a screening. A matched group of individuals without AAA will be included as control patients and followed with blood samples and questionnaires.

SUMMARY:
The number of AAA-surgeries performed per capita is 3-4 times higher in Innlandet county, as compared to Oslo. The last three years the annual incidence of AAA requiring treatment has been 21.5 / 100 000 inhabitants in Innlandet, as compared to 6.6 / 100 000 in Oslo. The indication for surgery is the same in both regions. In Oslo, a screening program was established in 2011, reporting a prevalence of AAA of 2.6 %, but in Innlandet county all AAA are either symptomatic or incidental findings and the prevalence is unknown. The aetiology of the major difference in AAA prevalence between these two regions has not been previously explored.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is a dilatation of the main artery from the heart as it passes through the abdomen. In case of rupture, the condition is life threatening and acute surgery is required. The prevalence of AAA is four to six times higher in men as compared to women, and varies greatly between countries and regions, but is generally reported to be present in 1.5-5% of men. Over the last three decades, the prevalence of AAA has been relatively stable, despite improved medical therapy for cardiovascular disease and a declining use of tobacco in Norway and comparable countries. This may in part be a consequence of unchanged aneurysmal progression rate combined with improved life expectancy of individuals at risk of developing AAA. Approximately 1% of all deaths in men over 65 years of age in Norway is caused by a ruptured AAA. The mortality is 75-80% after rupture, and half the patients die before they reach a hospital with vascular surgery. A patient with an incidental finding of AAA will be offered surgery in an elective setting to prevent rupture. The number of AAA surgeries in Norway was 851 in 2021 according to the Norwegian Vascular Surgery Registry (NORKAR).

The key challenge in improvement of aneurysm related mortality is to detect the disease while it is still asymptomatic. Screening is required to detect an asymptomatic AAA and is considered a beneficial healthcare intervention in several European countries.

We hypothesize that the prevalence of AAA is significantly higher in Innlandet, as compared to Oslo, and further, that the discrepancies in AAA prevalence between regions may be caused by differences in prevalence of risk factors, medication, socio-economic status, or in variations in genetic susceptibility.

Several genetic markers and other biomarkers have been proposed to relate to aneurysm disease. Of the clinically applicable biomarkers D-dimer, LDL cholesterol, HDL cholesterol, Thrombocytes, Apolipoprotein B and HbA1c have been found to have the most significant association to aneurysm growth rate. Studies on biomarkers for AAA have been hampered by low number of patients and currently no specific biomarker has been identified as a tool to identify patients with AAA or to predict aneurysm growth and studies on larger populations of patients with AAA have been called for.

The number of AAA-surgeries performed per capita is 3-4 times higher in Innlandet county, as compared to Oslo. The last three years the annual incidence of AAA requiring treatment has been 21.5 / 100 000 inhabitants in Innlandet, as compared to 6.6 / 100 000 in Oslo. The indication for surgery is the same in both regions. In Oslo, a screening program was established in 2011, reporting a prevalence of AAA of 2.6 %, but in Innlandet county all AAA are either symptomatic or incidental findings and the prevalence is unknown. The aetiology of the major difference in AAA prevalence between these two regions has not been previously explored.

There is some data on the psychological impact of a AAA screening and how a screening may impact the quality of life in patients diagnosed with AAA. However, there are still uncertainties towards the potential psychological harm of AAA screening, and further studies are required. Additionally, patients with AAA have in small studies an 80% reported prevalence of moderate to severe erectile dysfunction which is significantly higher than in the general population. Erectile dysfunction is also found to have an impact on the individual's quality of life, but the data on erectile dysfunction in AAA patients is limited.

Only men are included in the study. A prevalence of ≥1.5% is considered the cut-off for cost-benefit for screening for AAA. Previous studies have concluded that screening of women is not clinically indicated or cost-effective. Evaluation of recent data from the Norwegian Vascular Surgery registry has shown a stable proportion of women treated for AAA in Innlandet over several years. Consequently, women will not be incorporated into the study.

ELIGIBILITY:
Inclusion Criteria:

* All men in Inland Norway are invited

Exclusion Criteria:

* unwilling or unable to concent

Ages: 65 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Only men included
Study Population: All men in Innland Norway
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-05-09 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence | 3 years
  Prevalence of AAA is examined by screening of all 65 year old men in Innland, Norway during a period of three years. Screening is performed by ultrasound measurement of AP outer-outer diameter.
Etiology | 3 years
  Etiology of the anticipated high prevalence of AAA is explored through questionnaires and blood samples. Baseline charactereristics is to be compared to a different region in Norway with a similar screening project, and to be compared with control patients.

SECONDARY OUTCOMES:
Aneurysm related mortality | 6 years
  The norwegian cause of death registry will be consulted to find aneurysm related mortality in the region before, during and after introduction of the screening program.
All cause mortality | 6 years
  The norwegian cause of death registry will be consulted to find aneurysm related mortality and all cause mortality in the region before, during and after introduction of the screening program.
Prevalence of peripheral arterial insufficiency | 3 years
  Ankle brachial index will be measured in all patients. Ankle brachial index is a the measure of systolic blood pressure in the arm compared to the systolic blood pressure at the ankle. A normal ABI is 0,9-1,2, ranging from 0-1,5 (over 1,5 = incompressible vessels)
Prevalence of erectile dysfunction | 3 years
  Patients will be asked to fill out IIEF (erectile function questionnaire) to evaluate the prevalence and degree of erectile dysfunction in Inland Norway. 5 questions, each ranging from 1-5.
Quality of Life following screening | 6 years
  Effect of screening on qol are measured with SF-36 at baseline, 6 months and one year. A score from 0-100 is obtained through the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Simen T Berge, MD PhD, Study Chair — Sykehuset Innlandet, UiO; Chrissie M Andersen, MD, Principal Investigator — Sykehuset Innlandet, UiO
Locations (1):
- Sykehuset Innlandet, Hamar, Hamar, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Altreuther M. NORKAR Årsrapport for 2021 med plan for forbedringstiltak. St. Olavs Hospital; 2022.
- [Background] Lindholt JS, Diederichsen AC, Rasmussen LM, Frost L, Steffensen FH, Lambrechtsen J, Urbonaviciene G, Busk M, Egstrup K, Kristensen KL, Behr Andersen C, Sogaard R. Survival, Prevalence, Progression and Repair of Abdominal Aortic Aneurysms: Results from Three Randomised Controlled Screening Trials Over Three Decades. Clin Epidemiol. 2020 Jan 23;12:95-103. doi: 10.2147/CLEP.S238502. eCollection 2020. PMID 32158272
- [Background] Frønsdal KB, Svensjö S, Movik E, Desser AS, Smedslund G. Abdominalt aortaaneurisme (AAA) screening av menn i alder 65 år. 2020.
- [Background] Rabben T, Mansoor SM, Bay D, Sundhagen JO, Guevara C, Jorgensen JJ. Screening for Abdominal Aortic Aneurysms and Risk Factors in 65-Year-Old Men in Oslo, Norway. Vasc Health Risk Manag. 2021 Sep 10;17:561-570. doi: 10.2147/VHRM.S310358. eCollection 2021. PMID 34531660
- [Background] Ali MU, Fitzpatrick-Lewis D, Kenny M, Miller J, Raina P, Sherifali D. A systematic review of short-term vs long-term effectiveness of one-time abdominal aortic aneurysm screening in men with ultrasound. J Vasc Surg. 2018 Aug;68(2):612-623. doi: 10.1016/j.jvs.2018.03.411. PMID 30037679
- [Background] Nana P, Dakis K, Brodis A, Spanos K, Kouvelos G. Circulating Biomarkers for the Prediction of Abdominal Aortic Aneurysm Growth. J Clin Med. 2021 Apr 16;10(8):1718. doi: 10.3390/jcm10081718. PMID 33923412
- [Background] Lyttkens L, Wanhainen A, Svensjo S, Hultgren R, Bjorck M, Jangland E. Systematic Review and Meta-Analysis of Health Related Quality of Life and Reported Experiences in Patients With Abdominal Aortic Aneurysm Under Ultrasound Surveillance. Eur J Vasc Endovasc Surg. 2020 Mar;59(3):420-427. doi: 10.1016/j.ejvs.2019.07.021. Epub 2020 Jan 10. PMID 31928908
- [Background] Ericsson A, Kumlien C, Ching S, Carlson E, Molassiotis A. Impact on Quality of Life of Men with Screening-Detected Abdominal Aortic Aneurysms Attending Regular Follow ups: A Narrative Literature Review. Eur J Vasc Endovasc Surg. 2019 Apr;57(4):589-596. doi: 10.1016/j.ejvs.2018.10.012. Epub 2019 Mar 22. PMID 30910494
- [Background] Falkensammer J, Hakaim AG, Falkensammer CE, Broderick GA, Crook JE, Heckman MG, Oldenburg WA, Hugl B. Prevalence of erectile dysfunction in vascular surgery patients. Vasc Med. 2007 Feb;12(1):17-22. doi: 10.1177/1358863X06076043. PMID 17451089
- [Background] Elterman DS, Bhattacharyya SK, Mafilios M, Woodward E, Nitschelm K, Burnett AL. The Quality of Life and Economic Burden of Erectile Dysfunction. Res Rep Urol. 2021 Feb 18;13:79-86. doi: 10.2147/RRU.S283097. eCollection 2021. PMID 33634039
- [Background] Scott RA, Bridgewater SG, Ashton HA. Randomized clinical trial of screening for abdominal aortic aneurysm in women. Br J Surg. 2002 Mar;89(3):283-5. doi: 10.1046/j.0007-1323.2001.02014.x. PMID 11872050
- [Background] Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Pena BM. Development and evaluation of an abridged, 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res. 1999 Dec;11(6):319-26. doi: 10.1038/sj.ijir.3900472. PMID 10637462
- [Background] Bath MF, Sidloff D, Saratzis A, Bown MJ; UK Aneurysm Growth Study investigators. Impact of abdominal aortic aneurysm screening on quality of life. Br J Surg. 2018 Feb;105(3):203-208. doi: 10.1002/bjs.10721. PMID 29405273